CLINICAL TRIAL: NCT04940767
Title: A Prospective, Multicenter, Randomized, Evaluator-Blinded, Study to Evaluate the Safety and Efficacy of AMZEEQ® Companion Treatment With Oral Isotretinoin Therapy in Patients With Moderate to Severe Acne Vulgaris
Brief Title: A Companion Treatment Study for Patients With Moderate to Severe Acne Vulgaris
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Edward Lain, MD (Network)
Collaborators: Vyne Therapeutics Inc. (Industry)
Responsible Party: Sponsor-Investigator, Edward Lain, MD, Principal Investigator/Executive Director, Austin Institute for Clinical Research
Organization: Austin Institute for Clinical Research (Network)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: V77-123
Record Dates: First submitted 2021-06-16; First posted 2021-06-28 (Actual); Last update posted 2023-06-22 (Actual); Status verified 2023-06

CONDITIONS: Acne Vulgaris
MeSH Terms: conditions — Acne Vulgaris | interventions — Isotretinoin; Minocycline

STUDY DESIGN:
Who Masked: Investigator
Masking Description: Study evaluators will be blinded to patient treatment group allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Treatment Group A (Experimental): Patients will concomitantly receive once daily treatment of oral isotretinoin and topical AMZEEQ® for 20 weeks, followed by a further 24 weeks of once daily AMZEEQ® only treatment.
  Interventions: Drug: Isotretinoin; Drug: Amzeeq 4% Topical Foam
- Treatment Group B (Experimental): Patients will receive once daily treatment of oral isotretinoin for 20 weeks, followed by a further 24 weeks of once daily AMZEEQ® only treatment.
  Interventions: Drug: Isotretinoin; Drug: Amzeeq 4% Topical Foam

INTERVENTIONS:
Drug: Isotretinoin — Isotretinoin is a retinoic acid analogue (13-cis-retinoic acid) supplied as oral capsules. and was approved in the US for the treatment of severe acne vulgaris in 1982 under the brand name Accutane®.
  Other Names: Zenatane™
Drug: Amzeeq 4% Topical Foam — AMZEEQ® is a topical lipophilic foam containing 4% minocycline that was approved in the US for the treatment of acne vulgaris in 2019
  Other Names: minocycline

SUMMARY:
Acne vulgaris is a common disease of both males and females, usually manifesting initially during adolescence. The use of retinoic acid analogues such as adapalene, tazarotene and isotretinoin are also commonly prescribed to treat inflammation; dysregulated sebum production and comedonal acne. This study seeks to evaluate the efficacy and safety of concomitant use of both AMZEEQ® and oral isotretinoin compared to oral isotretinoin only use and to explore sequence dosing of both products as part of a long-term management protocol for acne vulgaris.

DETAILED DESCRIPTION:
Acne vulgaris is a common disease of both males and females, usually manifesting initially during adolescence. The primary pathologic events are initiated in the pilosebaceous units, especially of sebaceous-gland-bearing areas of the face, chest, and back as a result of increased androgen stimulation initiated at adrenarche or puberty. As a result of both abnormal keratinization of the infra-infundibular portion of the pilosebaceous follicle and increased sebum produced in the gland, a blockage of the duct results in the unapparent clinical lesion of the microcomedone. Continued blockage, colonization of the follicle by Cutibacterium acnes (C. acnes), and generation of multiple chemoattractant and proinflammatory moieties may result in non-inflammatory clinical lesions, comedones, and inflammatory lesions: papules, pustules, nodules, and cysts.

Acne treatments vary widely and frequently involve therapy combination approaches to achieve the objectives of initial disease control and long-term maintenance of effect. Antibiotics, especially clindamycin, minocycline, and doxycycline, have been prescribed as acne treatments for many years. These antibiotics effectively control the signs of inflammatory acne while patients continue to use them. Equally, the use of retinoic acid analogues such as adapalene, tazarotene and isotretinoin are also commonly prescribed to treat inflammation; dysregulated sebum production and comedonal acne.

AMZEEQ® is a topical lipophilic foam containing 4% minocycline that was approved in the US for the treatment of acne vulgaris in 2019 although minocycline containing products have been available in the US since the early 1970s. Minocycline is a semi-synthetic, second-generation tetracycline that imparts both a bacteriostatic and anti-inflammatory effect in the treatment of inflammatory acne. In addition, AMZEEQ® has been previously shown in clinical studies to positively impact comedonal acne.

Adverse events relating to oral minocycline use include tissue depigmentation primarily related to the ability of minocycline to complex with metals such as calcium and sequester into a variety of tissues e.g. bone, teeth and skin; CNS effects affecting the vestibular system e.g. dizziness, blurred vision and rare episodes of intracranial hypertension. Oral minocycline has also been implicated in rare but serious reactions such as anaphylaxis, erythema multiforme and DRESS syndrome. Interestingly, these findings do not appear to have much applicability to topically applied minocycline (as AMZEEQ®), likely due to significantly lower systemic exposure to minocycline when dosed by the topical route.

Isotretinoin is a retinoic acid analogue (13-cis-retinoic acid) supplied as oral capsules. and was approved in the US for the treatment of severe acne vulgaris in 1982 under the brand name Accutane®. Isotretinoin is the only therapy that impacts on all of the major aetiological factors implicated in acne. It achieves this by influencing cell-cycle progression, cellular differentiation, cell survival and apoptosis which results in a significant reduction in sebum production, influences comedogenesis, lowers surface and ductal C. acnes and has anti-inflammatory properties.

Although isotretinoin can ameliorate all four of the primary drivers of disease pathology, resulting in impressive clinical outcomes for severe and/or recalcitrant patients, the safety of isotretinoin continues to be a focal point for prescribers. As a teratogen, isotretinoin impacts the function of Hox genes that disrupts genetic control of axial patterning during embryo development. This can lead to developmental defects of the heart, spinal cord, palate, mandible, and other skeletal and neurological disorders such as hydrocephalus, microcephaly, and mental retardation. As such, careful monitoring of patients of both sexes via a risk evaluation and mitigation program (REMS) such as iPledge is a prerequisite for the safe use of the isotretinoin-containing products. Consequently, prescribers seek to discontinue oral isotretinoin use when it is appropriate to do so and to introduce other products with the goal of achieving a sustained long term clinical benefit for the patient.

The combination of these two, well-characterized acne treatments with two separate administration routes presents an intriguing, combined proposition of achieving rapid control of disease coupled with long-term disease management possibilities. As such this study seeks to evaluate the efficacy and safety of concomitant use of both AMZEEQ® and oral isotretinoin compared to oral isotretinoin only use and to explore sequence dosing of both products as part of a long-term management protocol for acne vulgaris.

ELIGIBILITY:
Inclusion Criteria:

Male or female patients will be considered eligible for participation in the study if all of the following inclusion criteria are satisfied prior to randomization:

1. Has completed and signed an appropriately administered Informed Consent Form (ICF) prior to any study-related procedures. Patients less than 18 years of age (or as required by state law) must sign an Assent Form for the study and a parent or legal guardian must sign the ICF.
2. Is 12 years of age or older.
3. Has facial acne vulgaris with an IGA score of moderate (3) or severe (4).
4. Is willing and able (with assistance from a caregiver as necessary) to both apply AMZEEQ® and take oral isotretinoin capsule(s) as directed, comply with study instructions, and commit to all follow-up visits for the duration of the study.
5. If female of child-bearing potential (FOCBP), must have two negative pregnancy tests, one being serologic, within the screening period.
6. Is willing to commit to true abstinence from heterosexual contact (which must be reviewed at each study visit and source documented) or agreed to use, and be able to comply with, effective contraception without interruption, prior to starting treatment as detailed below, during study period. For FOCBP who may participate in the study, the following methods of contraception, if properly used, are generally considered reliable with the following wait periods prior to having relations: oral contraceptives; vaginal contraceptive ring and patch contraceptives (one full cycle; e.g., 4 to 8 weeks); injection contraceptives (more than 7 days); intrauterine device or implantable hormone contraceptives (more than 7 days); surgical sterilization (bilateral tubal ligation) or a vasectomized partner (each, more than 6 months); male condom with intravaginal spermicide or diaphragm/cervical cap with spermicide (effective with proper use without a waiting period).
7. If sexually active male patient, must practice true abstinence (which must be reviewed at each study visit) or agree to use a condom with intravaginal spermicide during sexual contact with a pregnant female or a FOCBP, while participating in the study, during dose interruptions, and for at least 30 days following treatment discontinuation, unless patient has undergone a successful vasectomy. Male patients should refrain from making sperm donations at any time during study participation and for at least 30 days following treatment discontinuation.
8. Is willing to minimize exposure of the treated skin to ultraviolet light (e.g. avoid excessive sunlight, agree to not use tanning beds) and extremes in weather, such as wind or cold, throughout the study.
9. In the investigator's opinion, patient is in good general health and is free of any disease state or physical condition that exposes the patient to an unacceptable risk by study participation or impairs the evaluation of the patient or the treatments by participating in the study.

Exclusion Criteria:

Patients who meet any of the following will be excluded from the study:

1. Female who is pregnant, lactating or breastfeeding, or is planning a pregnancy during the study.
2. Acne conglobata, acne fulminans, secondary acne (chloracne, drug-induced acne), or any dermatological condition of the face (such as seborrhea, atopic dermatitis or basal cell carcinoma) that would require the use of confounding therapies or facial hair (eg, beard, sideburns, mustache) that could either interfere with clinical evaluations.
3. Sunburn on the face.
4. Severe systemic disease that might interfere with the conduct of the study or the interpretation of the results.
5. Abnormal Screening laboratory values that are considered clinically significant.
6. Patient is currently enrolled in another investigational drug or device study or is using or has used an investigational drug or investigational device treatment within 30 days of randomization.
7. Patient, who in the opinion of the investigator, is unable or unlikely to comply with the requirements of the study protocol.
8. Patients who have a history of any of the following will be excluded:

   * Allergy to tetracycline-class antibiotics or to any ingredient in the study drug
   * Pseudomembranous colitis or antibiotic-associated colitis
   * Hepatitis or liver damage or renal impairment
   * Known or suspected premalignant or malignant disease (excluding successfully treated skin cancers)
9. Patients who have used the following medications (topical refers only to the facial area) will not be eligible:

   * Within 1 week prior to randomization:

     * Medicated facial cleansers
     * Topical acne treatments (other than those listed below)
   * Within 4 weeks prior to randomization:

     * Topical retinoids on the face
     * Topical anti-inflammatories eg, PDE-4 inhibitors, calcineurin inhibitors and corticosteroids on the face
     * Topical corticosteroids on body areas other than the face for more than 15 consecutive days and on more than 10% of body surface area. In flexural body areas, such as axillary and inguinal regions, only mild topical corticosteroids and allowed for short term use (≤15 consecutive days).
     * Systemic antibiotics
     * Systemic acne treatments
   * Within 12 weeks prior to randomization:

     * Systemic retinoids
     * Systemic corticosteroids (Note: Intranasal and inhaled corticosteroids may be used throughout the study).
10. The following medications have been used less than the specified length of stable usage and patients must not initiate or change the dosing regimen during the course of the study: 3 months: hormonal contraceptives and therapies which also include testosterone replacement or supplementation.
11. Patient has any acute illness (eg, infection) within 48 hours of randomization, which, in the investigator's opinion, is considered significant.
12. Patient has a history of sensitivity to any of the ingredients in the medications.
13. Documented history of depression or self-harm that is not, in the opinion of the Investigator, currently adequately controlled with medication or in remission. Or, the presence of significant uncontrolled neuropsychiatric disorder, are clinically judged by the investigator to be at risk for suicide, or have a "yes" answer to any of the following at Screening or Baseline:

    1. Question 4 (Active Suicidal Ideation with Some Intent to Act, Without Specific Plan) on the "Suicidal Ideation" portion of the Columbia Suicide Severity Rating Scale (C-SSRS) or
    2. Question 5 (Active Suicidal Ideation with Specific Plan and Intent) on the "Suicidal Ideation" portion of the C-SSRS or
    3. Any of the suicide-related behaviors (actual attempt, interrupted attempt, aborted attempt, preparatory act or behavior) on the "Suicidal Behavior"portion of the C-SSRS.

    Note: A patient does not necessarily have to be excluded if they have self-injurious behavior that would be classified as non-suicidal self-injurious behavior. If this situation arises, the subject should be referred to a psychiatrist or appropriately trained professional as indicated.
14. Drug addiction or alcohol abuse (within the last 2 years).
15. Patient has history of previous use of isotretinoin.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2021-06-28 (Actual); Primary Completion 2023-04-28 (Actual); Study Completion 2023-04-28 (Actual)

PRIMARY OUTCOMES:
Lesion Improvement | 44 weeks
  Percent change from Baseline in inflammatory and comedonal lesion counts at each visit.
IGA Improvement | 44 weeks
  IGA Treatment Success (dichotomized as Yes/No) at each visit, where success is defined as an IGA score of 0 or 1, and at least a 2-grade improvement (decrease) from Baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Edward Lain, MD, MBA, Principal Investigator — Austin Institute for Clinical Research
Locations (2):
- United States (2):
  - Austin Institute for Clinical Research, Inc., Dripping Springs, Texas
  - Austin Institute for Clinical Research, Inc., Pflugerville, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Brown SK, Shalita AR. Acne vulgaris. Lancet. 1998 Jun 20;351(9119):1871-6. doi: 10.1016/S0140-6736(98)01046-0. No abstract available. PMID 9652685
- [Result] AMZEEQ® Prescribing Information - accessed March 10th 2021.
- [Result] Raoof TJ, Hooper D, Moore A, Zaiac M, Sullivan T, Kircik L, Lain E, Jankicevic J, Stuart I. Efficacy and safety of a novel topical minocycline foam for the treatment of moderate to severe acne vulgaris: A phase 3 study. J Am Acad Dermatol. 2020 Apr;82(4):832-837. doi: 10.1016/j.jaad.2019.05.078. Epub 2019 Jun 1. PMID 31163231
- [Result] Jones TM, Ellman H, deVries T. Pharmacokinetic Comparison of Once-Daily Topical Minocycline Foam 4% vs Oral Minocycline for Moderate-to-Severe Acne. J Drugs Dermatol. 2017 Oct 1;16(10):1022-1028. PMID 29036256
- [Result] Accutane® Prescribing Information - access March 10th 2021.
- [Result] Fogh K, Voorhees JJ, Astrom A. Expression, purification, and binding properties of human cellular retinoic acid-binding protein type I and type II. Arch Biochem Biophys. 1993 Feb 1;300(2):751-5. doi: 10.1006/abbi.1993.1104. PMID 8382035
- [Result] Allenby G, Bocquel MT, Saunders M, Kazmer S, Speck J, Rosenberger M, Lovey A, Kastner P, Grippo JF, Chambon P, et al. Retinoic acid receptors and retinoid X receptors: interactions with endogenous retinoic acids. Proc Natl Acad Sci U S A. 1993 Jan 1;90(1):30-4. doi: 10.1073/pnas.90.1.30. PMID 8380496
- [Result] Levin AA, Bosakowski T, Kazmer S, Grippo JF. 13-cis retinoic acid does not bind to retinoic acid receptors alpha, beta and gamma. Toxicologist. 1992; 12: 181.
- [Result] Ott F, Bollag W, Geiger JM. Oral 9-cis-retinoic acid versus 13-cis-retinoic acid in acne therapy. Dermatology. 1996;193(2):124-6. doi: 10.1159/000246226. PMID 8884148
- [Result] Geiger JM, Hommel L, Harms M, Saurat JH. Oral 13-cis retinoic acid is superior to 9-cis retinoic acid in sebosuppression in human beings. J Am Acad Dermatol. 1996 Mar;34(3):513-5. doi: 10.1016/s0190-9622(96)90462-4. No abstract available. PMID 8609271
- [Result] Tsukada M, Schroder M, Roos TC, Chandraratna RA, Reichert U, Merk HF, Orfanos CE, Zouboulis CC. 13-cis retinoic acid exerts its specific activity on human sebocytes through selective intracellular isomerization to all-trans retinoic acid and binding to retinoid acid receptors. J Invest Dermatol. 2000 Aug;115(2):321-7. doi: 10.1046/j.1523-1747.2000.00066.x. PMID 10951254
- [Result] Nelson AM, Gilliland KL, Cong Z, Thiboutot DM. 13-cis Retinoic acid induces apoptosis and cell cycle arrest in human SEB-1 sebocytes. J Invest Dermatol. 2006 Oct;126(10):2178-89. doi: 10.1038/sj.jid.5700289. Epub 2006 Mar 30. PMID 16575387
- [Result] Tantibanchachai C, Isotretinoin (Accutane) as a teratogen, Embryo Project Encyclopedia. 2014; ISSN: 1940-5030; http://embryo.asu.edu/handle/10776/8040
- See also: Tantibanchachai C, Isotretinoin (Accutane) as a teratogen, Embryo Project Encyclopedia. — http://embryo.asu.edu/handle/10776/8040